CLINICAL TRIAL: NCT03157232
Title: Rainbow DCI vs. R1-25 Sensor SpHb Sub-Range Performance Equivalence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR18695-TP14480
Record Dates: First submitted 2017-04-14; First posted 2017-05-17 (Actual); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Group (Experimental): All subjects are enrolled into the test group and all subjects received both the Rainbow DCI and R1-25 sensor.
  Interventions: Device: Rainbow DCI and R1-25 sensor

INTERVENTIONS:
Device: Rainbow DCI and R1-25 sensor — Noninvasive Measurement of SpHb

SUMMARY:
In this study, the concentration of hemoglobin was measured using noninvasive pulse oximeter sensors and compared against the hemoglobin measurement from the subject's blood sample under controlled conditions. Data collected in the study was in the sub-range of 11-17 g/dL in the device's 8-17 g/dL specification range.

The purpose of the study was to evaluate a change in the sensor component and to assess performance equivalence in the sub-range. The performance of non-invasive hemoglobin is not uniform across the accuracy range.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must understand and consent to be in the study.
* American Society of Anesthesiology Class 1 (Healthy subjects without any systemic disease at all).

Exclusion Criteria:

* Subjects who have any systemic disease at all.
* Subjects who do not understand the study and the risks.
* Smokers.
* Subjects who are pregnant.
* Subjects having either signs or history or peripheral ischemia. Others deemed ineligible by the clinical staff.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06-19 (Actual); Primary Completion 2009-06-29 (Actual); Study Completion 2009-06-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 18
Age, Customized [Number; unit: participants]
  26-65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Sub-Range Performance Equivalence of Rainbow DCI and R1-25 Sensors by ARMS Calculation
Description: Sub-range performance equivalence was determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter sensor to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value.In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from the pulse oximeter hemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of these differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours per subject
Measure: Number; unit: g/dL
Arm/Group | Test Group
Number analyzed (Participants) | 18
g/dL
  Rainbow DCI | 1.2
  R1-25 | 1.2

ADVERSE EVENTS:
Arm/Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes